CLINICAL TRIAL: NCT06655233
Title: Profiling the Intratumoral Microbiome of Pancreatic Ductal Adenocarcinoma Based on EUS-FNB Tissue Samples and Exploring Its Impact on Tumor Diagnosis and Prognosis.
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Tian, MD, Li Tian, MD [fu3tianli], The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli4
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer; EUS-FNB; Intratumoral Microbiota; Diagnosis; Prognosis
Keywords: pancreatic cancer; EUS-FNB; intratumoral microbiota; diagnosis; Prognosis
MeSH Terms: conditions — Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To minimize trauma for pancreatic disease patients and adhere to ethical requirements, we strictly use residual tissue from the EUS-FNB procedure for microbiome sequencing. During EUS-FNB, we first perform Rapid On-Site Evaluation (ROSE) to preliminarily assess sample quality and suitability. Based on quick pathological evaluation results, appropriate residual tissue is selected for microbiome analysis. This ensures sample quality and maximizes the use of residual tissue from clinical diagnostics, avoiding additional collection and meeting ethical standards. Patients undergo EUS-FNB based solely on clinical necessity, not for research purposes. The retained pancreatic tissue (about one strip) from EUS-FNB will be used for microbiome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to use endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) to investigate the intratumoral microbiome profile in patients with pancreatic ductal adenocarcinoma (PDAC) and to evaluate its potential impact on tumor diagnosis and prognosis. PDAC is the most common and lethal type of pancreatic cancer, accounting for over 85% of all pancreatic cancer cases. Given that most patients are diagnosed at an advanced stage when surgery is no longer an option, EUS-FNB serves as a crucial and minimally invasive method for accessing and analyzing the microbiome within the tumor.

The main questions this study aims to answer are:

Can EUS-FNB reliably and accurately detect the microbiome within PDAC tumors?

Researchers will analyze tissue samples obtained through EUS-FNB to confirm its ability to accurately capture the diversity and composition of the tumor microbiome.

Are there specific microbes or metabolites within the PDAC tumor microbiome that are linked to patient prognosis or response to chemotherapy?

The study will screen for and identify key microbial species or metabolites associated with treatment outcomes and patient survival in PDAC.

To ensure the reliability of the EUS-FNB results, researchers will systematically compare microbiome data obtained from EUS-FNB samples with those from surgical biopsies of pancreatic cancer tissue. This comparison will help validate the consistency and accuracy of the two methods in identifying the microbiome diversity and composition, confirming the clinical and research utility of EUS-FNB.

Participant Requirements:

Participants will be patients diagnosed with PDAC who require EUS-FNB as part of their clinical assessment and treatment pathway.

During the EUS-FNB procedure, researchers will use the remaining tissue after rapid on-site evaluation (ROSE) to conduct microbiome sequencing, ensuring sample quality.

All participants will provide informed consent, allowing the use of leftover tissue for microbiome analysis, and their privacy will be strictly protected throughout the study.

Study Procedures:

Participants will undergo a standard EUS-FNB procedure as part of their routine clinical care, with no additional procedures required for the study.

Researchers will compare the microbiome characteristics from EUS-FNB samples with those from surgical biopsy samples to verify consistency.

The study will utilize 2bRAD-M metagenomic sequencing technology, which is cost-effective and suitable for low-biomass, host-contaminated, and degraded microbiome samples. This method generates an accurate species-level taxonomic profile for analysis.

By identifying key microbial components or metabolites linked to patient prognosis or treatment response, this study aims to provide scientific evidence for early detection strategies and effective treatment plans for PDAC patients, potentially bringing significant clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 18 and 80 years.
2. Patients with pancreatic lesions confirmed through imaging examinations (US, MRI, CT, or PET-CT) with a high suspicion of pancreatic ductal adenocarcinoma (PDAC) who require EUS-FNB for diagnostic assistance.
3. Patients who have not received any chemotherapy, including neoadjuvant, postoperative adjuvant, or palliative chemotherapy.
4. Patients who agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Poor physical condition, including but not limited to hemoglobin ≤ 8.0 g/dl, severe cardiopulmonary insufficiency, etc.
2. Coagulation disorders (platelet count < 50 × 10^9/L, international normalized ratio > 1.5).
3. Failed anesthesia evaluation.
4. Acute pancreatitis within the past 2 weeks.
5. Pregnant or breastfeeding individuals.
6. Mental illness, drug addiction, or other conditions that may affect follow-up.
7. Patients who have received antibiotic treatment before the biopsy procedure or other conditions deemed unsuitable by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At the Third Xiangya Hospital of Central South University, patients with pancreatic diseases requiring diagnosis through EUS-FNB.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Differences in Microbiome Diversity and Abundance Between Pancreatic Ductal Adenocarcinoma (PDAC) and Non-Cancerous Tissues | 2 years
  Using 2bRAD-M metagenomic sequencing technology, the study measures and compares bacterial species, quantity, and diversity between PDAC and non-cancerous tissues. This analysis evaluates the relationship between these microbial characteristics and the occurrence and progression of PDAC, aiming to uncover the potential role of the microbiome in the disease process.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Hunan, Hunan, China

IPD SHARING:
Plan to Share IPD: No
There is not plan to make IPD avaliable